CLINICAL TRIAL: NCT04370886
Title: Recruit Blood Donors Via SMS With Different Contents During Epidemic of COVID-19
Brief Title: Recruit Blood Donors Via SMS During Epidemic of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Blood Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Recruit Blood Donors via SMS
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-04

CONDITIONS: Blood Donation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SMS with safty ensurance (Experimental): SMS content in this group will be about what blood services will do to ensure the safety of blood donors' life saving donation during 2019-nCoV epidemic
  Interventions: Behavioral: blood donation SMS
- SMS with saving life call-1 (Experimental): SMS content in this group will be about calling the blood donors to a life saving donation
  Interventions: Behavioral: blood donation SMS
- SMS with saving life call-2 (Experimental): SMS content in this group will be about calling the blood donors to a life saving donation
  Interventions: Behavioral: blood donation SMS
- SMS with holiday greeting (Placebo Comparator): SMS content in this group will be about holiday greeting of Labour Day.
  Interventions: Behavioral: blood donation SMS

INTERVENTIONS:
Behavioral: blood donation SMS — The literature shows that the information extraction and processing in emergency is different from the normal situation. To find the most effective emergency recruitment method during an outbreak, we intervened with a well-balanced group of donors by presenting different emergency recruitment text messages.

SUMMARY:
The fight against the spread of the 2019-nCoV epidemic has achieved some success in China, but the epidemic is far from over. A key factor making the epidemic under control in China is the government's call for social distance, which has led to few people going out for donation. As a result, the number of blood donors on the streets has been continuing to decline. Urgent recruitment of blood donors is therefore planned during the period from 30 April to 10 May via emergency recruitment SMS . This study has been designed to compare which information extraction frameworks would be more sensitive to blood donors in emergency situations.

DETAILED DESCRIPTION:
Researches has showed that that the information extraction and processing in emergency was different from the normal situation. To understand what information the blood donors are more sensitive to in an environment that may pose a potential threat to themselves, this interventional study has been designed. Eligible blood donors in Guangzhou Blood Center has been randomly divided into four groups according to their sociological variables, their interval since last blood donation , their history donation times and the location of their last blood donation. Three groups of donors has been randomly selected as interventional groups, and will receive three kindly of emergency blood donor recruitment SMS respectively. The placebo group donors will only receive a May Day greeting SMS.

One blood donor recruitment SMS will emphasize what blood services will do to ensure the safety of blood donors during their donation in 2019-nCoV epidemic, one will shows information about a loss-based framework, while the third one will show information about a benefit-based framework .

ELIGIBILITY:
Inclusion Criteria:

* blood donors whose last turning up were between October 31, 2016 to October 31, 2019

Exclusion Criteria:

* Blood donors who were deferral by blood screening result and other situations. Blood donors who have indicated that they would not accept urgent recruitment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 456517 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Blood donation rate | 10 days
  Blood donation rate of donors in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Blood Center, Guangzhou, Guangdong, China